CLINICAL TRIAL: NCT02433470
Title: Association of Functional Changes in the Brain and the Perception of Pain in Patients With Chronic Inflammatory Bowel Diseases (IBD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Magdalena S. Prüß née Volz, Dr. med. Magdalena Sarah Prüß (geb. Volz), Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EA4/028/15
Record Dates: First submitted 2015-04-25; First posted 2015-05-05 (Estimated); Last update posted 2018-01-24 (Actual); Status verified 2018-01

CONDITIONS: Inflammatory Bowel Disease
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- Active tDCS (Active Comparator): Active transcranial direct current stimulation
  Interventions: Device: Transcranial direct current stimulation
- Sham tDCS (Sham Comparator): Sham transcranial direct current stimulation
  Interventions: Device: Transcranial direct current stimulation

INTERVENTIONS:
Device: Transcranial direct current stimulation — Transcranial direct current stimulation over the motor cortex
  Other Names: tDCS

SUMMARY:
In the study the investigators aim to test whether transcranial direct current stimulation (tDCS)-induced pain reduction is in association with functional changes in the brain measured with magnetic resonance imaging (MRI) in patients with chronic inflammatory bowel diseases (IBD).

Hypothesis: Transcranial direct current stimulation can reduce the perception of pain in patients with chronic inflammatory bowel diseases, which is in association with changes in the brain measured via MRI.

ELIGIBILITY:
Inclusion Criteria:

* Inflammatory bowel disease
* Chronic pain (more than 3 months)
* Pain (VAS > 3/10)

Exclusion Criteria:

* Contraindication to transcranial direct current stimulation
* Contraindications to magnetic resonance imaging (MRI)
* Pregnancy
* Sever internal or psychiatric condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-04; Primary Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Functional and/or structural changes in the brain measured with cerebral MRI | 1 week
  Participants will be followed for 2 weeks
Changes in perception of pain measured with visual analogue scale and pain pressure threshold | 2 weeks
  Participants will be followed for 2 weeks

SECONDARY OUTCOMES:
Changes in quality of life | 2 weeks
Changes in functional symptoms (questionnaire: Irritable bowel syndrome - severity scoring system (IBS-SSS)) | 2 weeks
  Questionnaire: irritable bowel syndrome - severity scoring system (IBS-SSS)
Changes in activity indices (Harvey-Bradshaw Index (HBI) or simple clinical colitis activity index) | 2 weeks
  (Harvey-Bradshaw Index (HBI) or simple clinical colitis activity index)
Changes in pain catastophizing scale | 2 weeks
Changes in inflammation bBlood) | 2 weeks
Changes in inflammation (stool - calprotectin) | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Magdalena S Prüß-Volz, MD, Principal Investigator — Charite University
Locations (1):
- Charite University Medicine, Berlin, Germany